CLINICAL TRIAL: NCT05548036
Title: A Feasibility Randomised Control Trial (RCT) of Aerobika TM Verses Active Cycle of Breathing Technique (ACBT) in People With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Feasibility RCT of Aerobika Verses ACBT in People With COPD
Acronym: TIPTOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carwyn Bridges (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government); Trudell Medical International (Industry); Respiratory Innovation Wales (Unknown)
Responsible Party: Sponsor-Investigator, Carwyn Bridges, Hon research fellow, Hywel Dda Health Board
Organization: Hywel Dda Health Board (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/WA/0144
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: COPD; Bronchiolitis
Keywords: airways clearance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Masking Description: Randomised at recruitment then due to the nature of the intervention masking is not viable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPEP (Active Comparator): Oscillatory Positive Expiratory Pressure OPEP is a technique aimed at loosening and mobilising secretions it can be achieved by using a device (AerobikaTM). The device provides pulses of resistance as you exhale acting to open airways and shake secretions, enabling expectoration using a huff and cough technique. Key factors to consider when completing a treatment session are body position, users should be seated, with good posture, in a comfortable position.
  Interventions: Device: OPEP
- ACBT (Active Comparator): Active Cycle of Breathing Technique ACBT is a method of breathing performed in a cycle, used to help loosen and clear secretions from within the lungs (Panaligan et al., 2012). It consists of three different phases.
  Interventions: Device: OPEP

INTERVENTIONS:
Device: OPEP — OPEP (Aerobika (tm)
  Other Names: ACBT

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common preventable and treatable respiratory condition. Its main symptoms include, breathlessness, cough and frequent chest infections. Many people with COPD struggle with excessive production of sputum, resulting in more hospital admissions and worse symptoms affecting quality of life.

Guidelines suggest techniques to help clear sputum but there is not strong evidence behind these. In particular we don't know how effective cough clearance techniques are and indeed if any are better than others. This study will recruit people admitted to hospital with an exacerbation of COPD who have excessive sputum and randomise them to receive a hand-held airways clearance device or chest physiotherapy exercises. We will compare symptoms, quality of life, treatment burden and hospital admissions over the following year.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common, preventable and treatable disease and in the UK around 80% is caused by smoking. Respiratory symptoms include breathlessness, cough and excess sputum production. COPD is associated with significant healthcare burden and increased mortality and morbidity (GOLD, 2020).

Exacerbations are acute periods of worsening symptoms above normal day to day variation, leading to increased treatment and often emergency hospital admissions placing a significant burden on the health care system and are associated with a worse QoL and poorer long-term prognosis. (Ekberg-Aronsson et al., 2005). COPD causes over 30,000 deaths in the UK annually, and is the second commonest cause of hospital admission (NICE, 2018).

Patients with a chronic bronchitis phenotype have worse health status and COPD Assessment Test (CAT) score, experience more frequent exacerbations and received more pharmacological treatment than other phenotypes (Cosio et al., 2016).

Airways clearance appears an important adjunctive treatment in those with a chronic bronchitis phenotype of COPD who struggle with mucus hypersecretion (Svenningsen et al., 2016) but the evidence is not strong. In particular there are no well-designed studies (Randomised control trials-RCT's) that compare different types of cough clearance techniques against medication alone or against each other.

Burudpakdee et al. (2017) in a retrospective Canadian database analysis enrolled 405 participants into two crossmatch groups over a two-year period, found that provision of Oscillatory Positive Expiratory Pressure (OPEP) Aerobika™ devices were associated with a 19% re-exacerbation rate, compared with a 28% exacerbation rate in those receiving standard care (p=0.01). They suggested Aerobika™ may be a cost-effective way of reducing emergency department visits and costs associated with unplanned admissions. However, as this was a retrospective study, the data used to make these assumptions may lack clinical detail and be prone to reporting and selection bias.

The physiological rational for the use of AerobikaTM is demonstrated in Svenningsen et al. (2016) in a randomised crossover study. Regular use of Aerobika™ improved ventilation through sputum mobilisation which seemed to have a positive effect on QoL, ease of expectoration and pulmonary function -Forced Vital Capacity (FVC).

Several studies including Khoudigian-Sinani et al. (2017) and Thanh et al. (2019) analysed the cost effectiveness of the provision of an Aerobika™ in the United States and Canada respectively. Both studies concluded that Aerobika™ provided good value for money in reducing healthcare costs.

NICE (2018) guidelines state:

"If people have excessive sputum, they should be taught how to use positive expiratory pressure devices or active cycle of breathing techniques".

Despite a paucity of evidence NICE (2018) regard both OPEP (Aerobika™) and Active Cycle of Breathing Techniques (ACBT) as standard care in those people with COPD with excessive secretions. The reality in clinical care is that ACBT forms the first line treatment option with OPEP AerobikaTM offered as second line due to funding. There is a lack of evidence to support this decision making.

OBJECTIVES AND OUTCOME MEASURES/ENDPOINTS Rationale This study aims to provide some more robust information to inform clinicians of the effectiveness and tolerability of ACBT or OPEP (AerobikaTM) as part of an airway's clearance regime, in people with COPD and a chronic bronchitis phenotype.

5.2. Aims and Objectives A feasibility Randomised Control Trial (RCT) including real world evidence to assess the outcomes of OPEP (AerobikaTM) for people with COPD with a chronic bronchitis phenotype Primary Objectives

• To test the null hypothesis there is no difference in LCQ between groups at 3 months

Secondary Objectives

* To test the null hypothesis there is no difference in CAT between groups at 3 months
* To test the null hypothesis there is no difference in numbers and duration of hospital admissions at 1, 6 and 12 months.
* To compare numbers and duration of hospital admissions in the 12 months prior to starting the trial and 12 months after starting the trial within and between each group
* Time to first exacerbation between groups
* To compare number of courses of oral antibiotics or steroids
* To compare reported healthcare contacts in both groups at 1, 3 and 12 months
* To compare the proportions of participants achieving a change of >+2 on the LCQ in the ACBT versus OPEP groups at 3 and 12 months
* To compare the proportions of participants achieving a change of >-2 on the CAT in the ACBT versus OPEP groups at 3 and 12 months
* To note measures of cough severity (LCQ) and Quality of Life (QoL) (CAT and SF-36) within groups over time
* To note patient feedback on the tolerability and acceptability of AerobikaTM and ACBT (free text and Likert questions)
* To identify refusal, study completion and adherence

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital (current inpatient) or recent exacerbation treated in the community within 14 days with systemic steroids and/or antibiotics
* Male or Female, aged 40-90 years
* A diagnosis of COPD
* Greater than 10 pack year history
* FEV1 /FVC Ratio <0.70 at any time point in the last 5 years
* Regular sputum production (most days for at least 3 months)
* Prescribed optimal pharmacological treatment
* Able to provide informed consent
* CAT score >15

Exclusion Criteria:

* Contraindications to OPEP, recent hemoptysis or pneumothorax
* Unable to use OPEP (manual dexterity)
* Unstable cardiac conditions in the opinion of the clinical team
* Life expectancy less than 12 months.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
To test the null hypothesis there is no difference in Leister Cough Questionnaire between groups at 3 months | 3 months
  LCQ is a validated cough questionnaire. It consists of a 19-part questionnaire with a Likert scale scoring system between 1-7 measurements of physical, psychological, and social domains.

SECONDARY OUTCOMES:
To test the null hypothesis there is no difference in CAT between groups at 3 months | 3 months
  The CAT outcome measure is used in COPD research. Gupta et al. (2014) report good internal consistency (0.88-0.98), validity (p=>0.05) and responsiveness within exacerbations increasing scores by 4-5 points and rehabilitation decreasing scores by 2-3. we will measure the numerical change in score

CONTACTS AND LOCATIONS:
Locations (1):
- Mr Carwyn Bridges, Cardiff, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No